CLINICAL TRIAL: NCT04631770
Title: Mediastinal Lymph Node Dissection Versus Spared Mediastinal Lymph Node Dissection in Stage IA Non-small Cell Lung Cancer Presented as Ground-glass Nodules: Study Protocol of a Phase III, Randomized, Multi-center Trial (MELDSIG) in China
Brief Title: Mediastinal Lymph Node Dissection Versus Spared Mediastinal Lymph Node Dissection in Stage I GGN NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2020306
Record Dates: First submitted 2020-11-15; First posted 2020-11-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-05

CONDITIONS: Lung Neoplasms; Lymph Node Excision
Keywords: Non-small cell lung cancer; Mediastinal lymph node dissection; Ground-glass nodules
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediastinal lymph node dissection group (Experimental): A
  Interventions: Procedure: Systemic mediastinal lymph node dissection
- Spared mediastinal lymph node dissection group (Active Comparator): B
  Interventions: Procedure: Spared mediastinal lymph node dissection

INTERVENTIONS:
Procedure: Systemic mediastinal lymph node dissection — Systematic hilar and mediastinal lymph node dissection.
  Arms: Mediastinal lymph node dissection group
Procedure: Spared mediastinal lymph node dissection — Mediastinal lymph node is spared in this group.
  Arms: Spared mediastinal lymph node dissection group

SUMMARY:
Lung cancer is the leading cause of cancer related death worldwide. Lobectomy or sub-lobectomy with mediastinal lymph node dissection is the standard surgery. About 50% lung nodules are pure ground-glass or part-solid nodules. Non-solid nodules rarely develop mediastinal lymph node metastasis. The present study is a prospective, multicenter and randomized clinical trial, comparing the overall survival and disease-free survival of whether performing mediastinal lymph node dissection in non-small cell lung cancer with ground-glass nodule CT features.

DETAILED DESCRIPTION:
The study is a non-inferior statistical comparison, with 681 patients in each group. The anticipated enroll period is 3 years, followed by observation period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Thin-slice HRCT shows single GGN with C/T ≤ 0.5 and no lymph node metastasis;
* Clinical stage IA NSCLC (TNM 8th classification) diagnosed prior or in surgery;
* No history of malignancies within past 5 years or lung surgery;
* No anti-cancer treatment prior to surgery.

Exclusion Criteria:

* Simultaneous or metachronous (within the past 5 years) double cancers;
* Active bacterial or fungous infection;
* Interstitial pneumonitis, pulmonary fibrosis, or severe pulmonary emphysema;
* Systemic steroidal medication;
* Uncontrollable diabetes mellitus; (vi) Uncontrollable hypertension or history of severe heart disease, heart failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1362 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival is defined as days from randomization to death from any cause, and it was censored at the last day when the patient was alive.

SECONDARY OUTCOMES:
Relapse-free survival | 5 years
  RFS time is defined as days from randomization to relapse or death for any patient.
Proportion of local recurrence | 5 years
  Proportion of local recurrence in any kind of recurrences.
Duration of hospitalization | 1-60 days
  Duration of hospitalization around surgery.
Duration of chest drainage tube placement | 1-60 days
  Duration of chest drainage tube placement after surgery.
Operation time | 20-180 minutes.
  Time duration of surgery.
Blood loss | 1-60 days
  Blood loss during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfa Zhenfa, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Ethics review board of Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after publication of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the follow-up period of the study.

REFERENCES:
- [Derived] Li C, Ni Y, Liu C, Liu R, Zhang C, Song Z, Liu H, Jiang T, Zhang Z. Mediastinal lymph node dissection versus spared mediastinal lymph node dissection in stage IA non-small cell lung cancer presented as ground glass nodules: study protocol of a phase III, randomised, multicentre trial (MELDSIG) in China. BMJ Open. 2023 Oct 28;13(10):e075242. doi: 10.1136/bmjopen-2023-075242. PMID 37898488